CLINICAL TRIAL: NCT00639821
Title: Mucosal Gene Expression Defects in Patients With Inflammatory Bowel Disease Before and After First Infliximab Therapy
Brief Title: Mucosal Gene Expression Defects in IBD
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Principal Investigator, Paul Rutgeerts, MD, PhD, KU Leuven
Other Study IDs: Array study IBD 1
Record Dates: First submitted 2008-03-14; First posted 2008-03-20 (Estimated); Last update posted 2012-10-22 (Estimated); Status verified 2012-10

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Gene expression microarray; Inflammatory bowel disease; Infliximab
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Ileal/colonic mucosal biopsies from patiens with inflammatory bowel disease refractory to corticosteroids and/or immunosuppression and from 12 control individuals
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- inflammatory bowel disease: Patients with refractory inflammatory bowel disease (ulcerative colitis and Crohn's disease) before and after treatment with infliximab.

SUMMARY:
This study investigated the mucosal gene expression defects associated with active Crohn's disease (CD)and ulcerative colitis (UC), and studied the effect of infliximab induced downregulation of inflammation and mucosal healing on these abnormalities, using whole genome gene expression microarrays.

DETAILED DESCRIPTION:
Infliximab, a monoclonal IgG1 antibody to the pro-inflammatory cytokine tumor necrosis factor-alpha (TNF-α), was the first efficacious biological therapy for IBD. Infliximab dramatically improved the quality of life in IBD patients. Besides inducing and maintaining remission in refractory IBD patients, infliximab has achieved new treatment goals such as intestinal mucosal healing and a reduction in hospitalizations and surgeries on the long-term. However, up to 30% of IBD patients do not respond to this costly therapy and potentially harmful therapy, and in an extra 20-30% response is incomplete. The mechanism of resistance to infliximab is unknown and predictors of response to infliximab are currently lacking.

The aim of this study was to investigate the mucosal gene expression defects associated with active Crohn's disease (CD)and ulcerative colitis (UC), and to study the effect of infliximab induced downregulation of inflammation and mucosal healing on these abnormalities, using whole genome gene expression microarray technology on endoscopic-derived intestinal mucosal biopsies from control individuals and patients with active IBD, and this before and after their first infliximab treatment.

Sixty-one patients with inflammatory bowel disease, 19 with Crohn's colitis, 18 with Crohn's ileitis and 24 with UC, undergo a colonoscopy with biopsies before and 4-6 weeks after the first infliximab treatment. Response to infliximab was defined based on endoscopic and histologic findings. A control group of 12 individuals was also included.Total RNA was isolated from biopsies, labelled and hybridized to Affymetrix HGU133plus2.0 Array. Microarray data were analyzed using Bioconductor software and Ingenuity Pathway Analysis software. Quantitative real time RT-PCR and immunohistochemistry were used to confirm microarray data.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Patients with inflammatory bowel disease refractory to corticosteroids and/or immunosuppression who had never been treated with biological therapy (anti-TNF treatment).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Colonic mucosal biopsies from patients with refractory inflammatory bowel disease who had never been treated with biological therapy.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2004-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Gene expression profiles assessed with microarray | before and after infliximab treatment (4-6 wks)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Rutgeerts, MD, PhD, Study Director — University of Leuven
Locations (1):
- Department of Gastroenterology, Leuven, Belgium

REFERENCES:
- [Derived] Arijs I, Li K, Toedter G, Quintens R, Van Lommel L, Van Steen K, Leemans P, De Hertogh G, Lemaire K, Ferrante M, Schnitzler F, Thorrez L, Ma K, Song XY, Marano C, Van Assche G, Vermeire S, Geboes K, Schuit F, Baribaud F, Rutgeerts P. Mucosal gene signatures to predict response to infliximab in patients with ulcerative colitis. Gut. 2009 Dec;58(12):1612-9. doi: 10.1136/gut.2009.178665. Epub 2009 Aug 20. PMID 19700435